CLINICAL TRIAL: NCT05147961
Title: Precision Medicine for Preventing Type 2 Diabetes: a Step Forward (PRE-MED2)
Brief Title: Precision Medicine for Preventing Type 2 Diabetes: a Step Forward
Acronym: PRE-MED2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Pisa (Other)
Collaborators: University of Florence (Other); Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Prof. Stefano Del Prato, Principal Investigator, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: University of Pisa _ Diabetes
Record Dates: First submitted 2021-09-13; First posted 2021-12-07 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: PreDiabetes
Keywords: Prediabetes; Diabetes prevention; Precision medicine; Circulating miRNA; Wereable device; Data integration; Obesity; Gestational Diabetes; Personalized risk estimation; mHealth
MeSH Terms: conditions — Prediabetic State; Obesity; Diabetes, Gestational | interventions — Digital Health; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth (Experimental): A mHealth automated behavioral intervention via E-mail, web, and mobile phone will be developed and tested in the intervention trial trial (phase 4 of the project)
  Interventions: Other: Digital Health
- Standard care (Active Comparator): Traditional recommendations (lifestyle modification) (phase 4 of the project)
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Digital Health — Automated behavioral intervention via e-mail, web, and mobile phone
  Arms: mHealth
Other: Standard care — Conventional recommendations on diet and exercise
  Arms: Standard care

SUMMARY:
The prevalence of type 2 diabetes (T2D) has been rising rapidly with an increased burden to the healthcare system. As such T2D prevention is highly recommendable, and, theoretically, it can definitely be successful. However, though feasible T2D prevention is difficult to implement due to the heterogeneity of the disease that make response to population intervention (and treatment) only partially successful. Precision medicine aims to prevent chronic diseases by tailoring interventions or recommendations to a combination of a genetic background, metabolic profile, and lifestyle. Classification of individuals at risk into clusters that differ in their susceptibility to develop T2D may foster the identification of preventive interventions. Recent advances in omics technologies have offered opportunities as well as challenges in the use of precision medicine to prevent T2D. Moreover, new mobile health (mHealth) technologies have enhanced how diabetes is managed. However, little is still known about the effectiveness of mHealth technology as intervention tools for reducing diabetes risk.

DETAILED DESCRIPTION:
Multicenter, interventional study (mHealth automated behavioral intervention versus traditional recommendations) designed: 1. toexplore the potential of more accurate subgroup distinction in prediabetes that may help to deliver a more effective preventive strategy with the final goal to enhance the possibility to prevent or delay the development of type 2 diabetes; 2. toexplore the use of mHealth to modify lifestyle in a subgroup of subjects known for their elevated risk of developing type 2 diabetes (i.e. obese and women with previous gestational diabetes) and to determine the impact of such strategies on the basis of individual characterization.

Phase 1: 1200 subjects at high risk of developing type 2 diabetes will be enrolled based on an opportunistic approach (FINDRISK questionnaire).The questionnaire will be made available at GP's offices, Pharmacies as well as through media.Moreover, the infrastructure for data collection and patient interventions will be developed.

Phase 2: all individuals will be characterized on the basis of diet habits (EPIC questionnaire; Binge Eating Scale) and physical activity (by a wrist-worn wearable device) as well metabolic profile (complete blood count, creatinine, plasma glucose and insulin, HbA1c, liver function tests, total cholesterol, HDL cholesterol, triglycerides, urine test, auto-antibody anti-GAD, and A/C ratio on urine spot sample; 75-g oral glucose tolerance test; HOMA-B and HOMA-IR)for identification of special subgroups.Circulating RNA and miRNAwill be extracted from lymphocytes and plasmafor identification ofbiomarkers for prediction of risk of disease and new targets for preventive intervention. A biobank of serum, urine and stool samples will be also collected genetic characterization and for omics profiling.

Phase 3, all lab determination and cluster analysis will be performed. All data will be integrated in the infrastructurefor the identification of new relevant factors and indicators useful for better understanding health conditions and outcomesand for the analysis of discrete risk subtypes (cluster).

Phase 4: the validity of themHealth approach on the metabolic and lifestyle attitude as a function of the individual characterization as obtained in Phase 3 will be tested in the exploratory clinical trial.ThemHealth automated behavioral intervention via E-mail, web, and mobile phone will be developed and tested in a trial in two high-risk populations of obese non-diabetic subjects (n=150) and women with previous gestational diabetes (n=150). These subjects will be randomized 1:1 to either 9-month conventional recommendation for correct lifestyle based on the procedures described in the Diabetes Prevention Programme or mHealth automated behavioral intervention via E-mail, web, and mobile phone. Subjects will be seen at 3-month interval for recording of anthropometric measurements and determination of fasting plasma insulin and glucose as well as lipid profile. During the last two weeks of the intervention trial all subjects will be provided with the same wearable device used for initial characterization for recording of the same initial parameters. At completion of the follow-up all initial measurements will be repeated.Data will then be analyzed as changes vs. baselines between the two groups as well as according to any sub-group.

ELIGIBILITY:
Inclusion Criteria:

* age of 18-70 years
* 12 points or more in the Finnish diabetes risk score or previous gestational diabetes or obese subjects
* technology skills (computers, smartphones, tablets with internet connection)
* absence of language barriers
* ability to provide written informed consent to the study

Exclusion Criteria:

* Established diagnosis of diabetes
* Pregnancy and breastfeeding
* Renal or hepatic failure
* Severe cardiovascular, neurological, hematological, endocrinological, gastrointestinal, nephrological or pneumological affections that may interfere with the study
* Ongoing treatment with antidiabetics, diuretics, glucocorticoids, antypsychoticsoral contraceptives or other drugs known to affect glucose metabolism.
* History of pancreatitis
* Alcohol abuse or abuse of psychoactive substances
* Subjects with mental disorders, or predictably unfit to understand and issue valid written informed consent to the study
* Subjects with mental disorders, or not suitable for understanding and performing the tasks required by the study
* Bariatric surgery
* Current cancer or less than 6 months from the end of cancer treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Development of type 2 diabetes, diagnosed by fasting or post-challenge plasma glucose concentrations meeting the American Diabetes Association criteria. | 9 months
  Number of subjects with a fasting glycemia ≥ 126 mg/dl or 2-h glycemia ≥200 mg/dl after ingestion of 75-g oral glucose load

SECONDARY OUTCOMES:
Economic evaluation | 9 months
  Cost-effectiveness of mHealth as compared to traditional approach for implementation of preventive measures
Identification of clustering by a machine learning approach | 9 months
  Rate of subjects with a different risk factor to develop type 2 diabetes identified by splitting the collected data by a machine learning algorithms
Identification of abnormal microbiome and metabolome | 9 months
  Number of subjects with abnormal microbiome and metabolome evaluated using sample type, feces, and others biosamples, such as urine, plasma/serum and analyzed by by reverse-phase ultra-high performance liquid chromatography-tandem mass spectrometry.
Bioinformatics and systems biology methodologies | 9 months
  Number of subjects estimated at risk of type 2 diabetes on the basis of the genomic profiles of the individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Del Prato, MD, Principal Investigator — Università di Pisa
Locations (2):
- Italy (2):
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - Stefano Del Prato, Pisa

IPD SHARING:
Plan to Share IPD: No